CLINICAL TRIAL: NCT06691061
Title: Real-life Comparative Effectiveness of Vedolizumab, Ustekinumab and JAK Inhibitors in Patients with Ulcerative Colitis After Anti-TNFα Failure or Intolerance
Brief Title: The PODIUM Study - a Three-arm Comparison of Target Therapies After Anti-TNFα in Ulcerative Colitis
Status: Recruiting | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Alessandro Armuzzi, Professor, Humanitas Clinical and Research Center
Other Study IDs: IBD-001-2023
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis (Disorder)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; Janus Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Vedolizumab — UC patients treated with vedolizumab
Drug: Ustekinumab - Standard Dosage — UC patients treated with ustekinumab
Drug: JAK Inhibitor — UC patients treated with JAK inhibitors

SUMMARY:
The goal of this observational study is to compare the real-life effectiveness and safety of vedolizumab, ustekinumab and JAK inhibitors in patients with UC who had been exposed to at least one anti-TNF-alpha therapy.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of UC according to the current European Crohn's and Colitis Organization (ECCO) guidelines7;
* Age ≥ 18 years-old;
* Capability of expressing informed consent;
* Clinically active ulcerative colitis (cf. 'operative clinical measures', below) at baseline;
* Initiation of vedolizumab, ustekinumab or JAK inhibitors (tofacitinib, upadacitinib or filgotinib) as second-line target therapy at baseline;
* Previous treatment with at least one anti-TNFα drug licenced for the treatment of UC (i.e., infliximab, adalimumab and/or golimumab);
* No exposure to vedolizumab, ustekinumab and JAK inhibitors before baseline;
* At least 1 follow-up visit after baseline

Exclusion Criteria:

* Diagnosis of Crohn's colitis, IBD-U or other gastrointestinal inflammatory conditions;
* Age < 18 years-old;
* Incapability of expressing informed consent;
* Acute severe UC requiring hospitalization at baseline;
* No previous exposure to anti-TNFα therapies;
* Previous treatment with target therapies other than anti-TNF-α for UC before baseline;
* Ustekinumab or JAK inhibitors induction with a non-standard posology for UC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and endoscopic effectiveness of the three treatments | 12 months
  Rates of steroid-free clinical remission and endoscopic remission

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital IRCSS, Mialn, Italy, Italy